CLINICAL TRIAL: NCT00831987
Title: Annual Study of Safety and Immunogenicity of Influenza Virus Vaccine Fluzone® 2004-2005
Brief Title: Safety and Immunogenicity of the World Health Organization (WHO) Formulation of the 2004-2005 Fluzone® Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC20
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2009-08-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Fluzone®; Influenza; Adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone® Vaccine Group - Age 18-59 Years (Experimental): Participants aged 18 to 59 years at enrollment and received 1 dose of Fluzone® Vaccine
  Interventions: Biological: Fluzone®: Influenza virus vaccine 2004-2005 formulation
- Fluzone® Vaccine Group - Age ≥ 60 Years (Experimental): Participants aged at least 60 years or older at enrollment and received 1 dose of Fluzone® Vaccine
  Interventions: Biological: Fluzone®: Influenza virus vaccine 2004-2005 formulation

INTERVENTIONS:
Biological: Fluzone®: Influenza virus vaccine 2004-2005 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone® Vaccine Group - Age 18-59 Years
Biological: Fluzone®: Influenza virus vaccine 2004-2005 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone® Vaccine Group - Age ≥ 60 Years

SUMMARY:
To observe and to describe the safety during Days 0 to 21 following injection of the 2004-2005 formulation of the inactivated, split-virion influenza vaccine Fluzone® in subjects aged 18-59 years and subjects aged ≥ 60 years.

To measure and to describe the immune response (antibodies to hemagglutinin) 21 days following injection of the 2004-2005 formulation of the inactivated, split-virion influenza vaccine Fluzone®, in subjects aged 18-59 years and subjects aged ≥ 60 years.

DETAILED DESCRIPTION:
The time of onset and duration of local and systemic solicited reactions will be assessed and reported. Unsolicited adverse events (including serious adverse events) will be collected and categorized throughout the study period.

Antibody levels will be evaluated by hemagglutination inhibition (HI) assay from sera obtained pre-vaccination (Day 0) and 21 days post-vaccination, for antigens from the 2004-2005 influenza virus strains: A/New Caledonia/20/99 (H1N1), A/Wyoming/03/2003 (H3N2), and B/Jiangsu/10/2003.

ELIGIBILITY:
Inclusion Criteria :

* Participant aged 18 years or older.
* Participant able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Participant is in reasonably good health as assessed by the investigator.
* Participant willing and able to meet protocol requirements.
* Participant willing and able to give informed consent.

Exclusion Criteria :

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever (temperature >100.4°F) in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature >100.4°F) on review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 3.
* Participation in any other experimental drug or vaccine trial within the 30 days preceding enrollment into the study.
* Immunogenicity or immunosuppressive therapy (including systemic steroid use for 2 weeks or more), cancer chemotherapy, or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past 3 months.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes mellitus requiring pharmacological control.
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing age, a positive urine pregnancy test, breast feeding, or not using a medically approved and reliable form of contraception (oral contraceptives or double barrier method) for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 06 through 16 August 2004 in 1 US site.
Pre-assignment Details: A total of 120 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone® Vaccine Group - Age 18-59 Years; Fluzone® Vaccine Group - Age ≥ 60 Years: Participants received 1 dose of Fluzone® vaccine on Day 0.
Period: Overall Study
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 4 | 64
  >=65 years | 0 | 56 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (11.1) | 74 (5.9) | 57.7 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 16 | 22 | 38
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local and Systemic Reactions After Fluzone® Vaccination
Description: Solicited local reactions: Erythema (redness), Induration, Bruising, and Pain at the injection site.
  Solicited systemic events: Fever (temperature), Chills, Rash, Headache, Cough, Runny nose, Nausea, Vomiting, Diarrhea, Malaise, Myalgia, and Arthralgia
Time Frame: 0 to 3 days post-vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Number analyzed (Participants) | 60 | 60
Percentage of Participants
  Any Solicited Local (Injection Site) Reaction | 60 | 23
  Any Erythema (> 0.5 cm) | 8 | 5
  Grade 3 Erythema (≥ 5.0 cm) | 0 | 2
  Any Induration (> 0.5 cm) | 7 | 0
  Grade 3 Induration (≥ 5.0 cm) | 2 | 0
  Any Bruising (> 0.5 cm) | 2 | 0
  Grade 3 Bruising (≥ 5.0 cm) | 0 | 0
  Any Pain | 60 | 20
  Grade 3 Pain (unable to perform usual activities) | 0 | 0
  Any Solicited Systemic Reaction | 42 | 23
  Any Fever (≥ 100.4 º F) | 0 | 0
  Grade 3 Fever (≥ 104.0 º F) | 0 | 0
  Any Headache | 23 | 8
  Grade 3 Headache (prevents daily activity) | 0 | 0
  Any Chills | 2 | 2
  Grade 3 Chills (prevents daily activity) | 0 | 0
  Any Cough | 7 | 3
  Grade 3 Cough (prevents daily activity) | 0 | 0
  Any Runny Nose | 8 | 3
  Grade 3 Runny Nose (prevents daily activity) | 0 | 0
  Any Rash | 0 | 0
  Grade 3 Rash (prevents daily activity) | 0 | 0
  Any Malaise | 7 | 2
  Grade 3 Malaise (prevents daily activity) | 0 | 0
  Any Myalgia | 13 | 8
  Grade 3 Myalgia (prevents daily activity) | 0 | 0
  Any Arthralgia | 7 | 2
  Grade 3 Arthralgia (prevents daily activity) | 0 | 0
  Any Nausea | 8 | 2
  Grade 3 Nausea (prevents daily activity) | 0 | 0
  Any Vomiting | 2 | 0
  Grade 3 Vomiting (≥ 3 per day) | 0 | 0
  Any Diarrhea | 3 | 5
  Grade 3 Diarrhea (≥ 5 episodes per day) | 0 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Antibodies Pre- and Post-Vaccination With Fluzone® Vaccine
Description: GMTs and their 95% Confidence Intervals for each of the 3 antigens pre- and post-vaccination with Fluzone® 2004-2005 formulation.
Time Frame: Day 0 and Day 21 Post-Vaccination
Population: Geometric Mean Titers were assessed in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Number analyzed (Participants) | 60 | 60
Titers
  A/NEW CALEDONIA/20/99 (H1N1) Pre-vaccination | 21.3 [15.7 to 28.9] | 15.6 [13.1 to 18.6]
  A/New CALEDONIA/20/99 (H1N1) Post-vaccination | 39.3 [29.0 to 53.3] | 19.8 [16.0 to 24.3]
  A/WYOMING/03/2003 (H3N2) Pre-vaccination | 34.2 [24.1 to 48.7] | 25.6 [20.1 to 32.6]
  A/WYOMING/03/2003 (H3N2) Post-vaccination | 85.7 [64.8 to 113.4] | 64.2 [46.2 to 89.1]
  B/JIANGSU/10/2003 Pre-vaccination | 8.5 [7.2 to 10.0] | 10.6 [9.1 to 12.4]
  B/JIANGSU/10/2003 Pre-vaccination | 23.5 [18.3 to 30.2] | 21.5 [16.3 to 28.5]

3. Primary Outcome: Percentage of Participants With at Least 40 Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination
Time Frame: 21 Days post-vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Number analyzed (Participants) | 60 | 60
Percentage of Participants
  A/NEW CALEDONIA/20/99 (H1N1) | 60 | 23
  A/WYOMING/55/2004 (H3N2) | 87 | 78
  B/JIANGSU/10/2003 | 45 | 33

4. Primary Outcome: Percentage of Participants With at Least a 4-Fold Increase in Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination
Time Frame: Day 21 post-vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Number analyzed (Participants) | 60 | 60
Percentage of Participants
  A/NEW CALEDONIA/20/99 (H1N1) | 18 | 5
  A/WYOMING/55/2004 (H3N2) | 35 | 33
  B/JIANGSU/10/2003 | 47 | 23

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 21 days post-vaccination.
Arm/Group | Fluzone® Vaccine Group - Age 18-59 Years | Fluzone® Vaccine Group - Age ≥ 60 Years
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 60/60 | 20/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine Group - Age 18-59 Years (N=60) | Fluzone® Vaccine Group - Age ≥ 60 Years (N=60)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone® Vaccine Group - Age 18-59 Years (N=60) | Fluzone® Vaccine Group - Age ≥ 60 Years (N=60)
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Injection site erythema (General disorders) | 8 | 5
Injection site induration (General disorders) | 7 | 0
Injection site pain (General disorders) | 60 | 20
Malaise (General disorders) | 7 | 2
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 8 | 2
Headache (Nervous system disorders) | 23 | 8
Headache (Nervous system disorders) | 10 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Rhinorrhoea (Runny nose) (Respiratory, thoracic and mediastinal disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications